CLINICAL TRIAL: NCT00248027
Title: Tracking Service Use and Outcomes II:First Episode Psychosis and Psychotic Disorders Clinic
Status: Terminated | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Other Study IDs: REB #04-203
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Schizophreniform,First Episode Psychosis
Keywords: early intervention,program evaluation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Main Research questions:

1. Who are the patients referred for treatment at the Psychotic Disorders Clinic?
2. What are the outcomes from treatment for first episode psychosis in multiple outcome domains?
3. What hospital resources are used over the early course of the illness?
4. How satisfied are patients and family with the treatment and services they received? This is an important study that will help us evaluate the service and treatment offered by the Psychotic Disorders Clinic's specialized early intervention program,which helps young people experiencing early stages of psychotic illness.A growing body of evidence suggests that intervening earlier in the course of the illness with specialized and complimentary pharmacological and psychosocial treatment may be associated with improved outcomes.

DETAILED DESCRIPTION:
The project is primarily a descriptive study of individuals experiencing their first episode of psychosis presenting at the Psychotic Disorders Clinic/Early Intervention Program.

The objectives of the study are:

1. Track multi-dimensional outcomes within the program
2. Track service use
3. Compare outcomes for this early intervention program with outcomes noted in published follow up studies
4. Evaluate effectiveness of the Psychotic Disorders Clinic in improving outcomes for persons experiencing their first episode of psychosis

ELIGIBILITY:
Inclusion Criteria:

* male or female between ages of 16 to 50 years of age
* capable of providing informed consent
* receiving treatment voluntarily
* experiencing a "first episode of psychosis" defined as the first episode of illness and where the subject,at presentation,meets DSM-IV criteria for one of the following diagnoses:schizophrenia,schizophreniform disorder,schizoaffective disorder,brief psychotic disorder,delusional disorder,and psychosis NOS

Exclusion Criteria:

* primary diagnosis of mood disorder
* diagnosis of substance-induced psychosis
* diagnosis of psychosis due to a general medical condition
* diagnosis of mental retardation
* diagnosis of developmental disorder
* has received antipsychotic treatment for greater than 1 month
* has received treatment for an earlier episode of psychosis from which there has been a remission of symptoms for greater than 3 months

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Archie, MD,FRCP(C), Principal Investigator — Assistant Professor Dept of Psychiatry and Behavioural Neurosciences McMaster University.Active Medical Staff Hamilton Health Sciences.Clinical Director of Cleghorn Early Intervention in Psychosis Program and Psychotic Disorders Clinic
Locations (1):
- Cleghorn Program-Early Intervention in Psychosis.St Joseph's Healthcare Hamilton/Hamilton Health Sciences, Hamilton, Ontario, Canada